CLINICAL TRIAL: NCT05686395
Title: Comparative Study of Analgesic Efficacy of Ultrasound Guided Interscalene Block Versus Combined Shoulder Anterior Capsular Block and Suprascapular Nerve Block for Arthroscopic Shoulder Surgeries.
Brief Title: Pain Control After Arthroscopic Shoulder Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hosameldin Ibrahim Ibrahim Elsayed Eldib, ASSISTANT LECTURER OF ANESTHESIA AND INTENSIVE CARE AND PAIN MEDICINE, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB0010038
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 Ultrasound-guided Interscalene Block group (Active Comparator): In this group, ultrasound-guided ISB will be done using 10 ml of bupivacaine 0.25%.
  Interventions: Procedure: Ultrasound-guided Interscalene Block group; Drug: Bupivacaine
- group 2 Combined Ultrasound guided shoulder anterior capsular block and suprascapular nerve block (Active Comparator): , ultrasound-guided SHAC block will be done using 10 ml of bupivacaine 0.25% injected in the interfacial plane between deltoid and subscapular muscle and 10 ml of bupivacaine 0.25% injected in the pericapsular space. Ultrasound-guided SSN block will be done using 10 ml of bupivacaine 0.25% injected at sub omohyoid space.
  Interventions: Procedure: Combined Ultrasound guided shoulder anterior capsular block and suprascapular nerve block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Ultrasound-guided Interscalene Block group — ultrasound guided interscalene block versus combined ultrasound guided shoulder anterior capsular block and suprascapular nerve block for arthroscopic shoulder surgery
  Arms: group 1 Ultrasound-guided Interscalene Block group
Procedure: Combined Ultrasound guided shoulder anterior capsular block and suprascapular nerve block — Combined Ultrasound guided shoulder anterior capsular block and suprascapular nerve block
  Arms: group 2 Combined Ultrasound guided shoulder anterior capsular block and suprascapular nerve block
Drug: Bupivacaine — bupivacaine 0.25%.

SUMMARY:
This study will be conducted to compare the perioperative analgesic efficacy of ultrasound - guided interscalene brachial plexus block versus combined shoulder anterior capsular block and anterior suprascapular nerve block for arthroscopic shoulder surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-65 years of both sexes, with American Society of Anesthesiologists (ASA) physical status I or II admitted for arthroscopic shoulder surgery.

Exclusion Criteria:

* Patient refusal.
* Uncooperative patient.
* Patient with neurological deficit.
* Patients with respiratory disorders.
* Patient with bleeding disorders.
* Infection at the block injection site.
* Patients with history of allergy to local anesthetics.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
post operative analgesic consumption | 24 hours after surgery
  The first 24 hours post operative analgesic consumption

SECONDARY OUTCOMES:
Visual Analogue score (VAS) in the first 24 hours after surgery | first 24 hours after surgery
  - Postoperative pain intensity will be assessed in the first 24 hour using VAS score where (0 = no pain and 100 = the worst imaginable pain)
Patient satisfaction score | first 24 hours after surgery
  Patient satisfaction score will be assessed on the basis of a questionnaire and graded on a 4-point scale (excellent/good/fair/poor).
The incidence of hemi diaphragmatic paralysis | immediately before block and immediately after procedure
  hemidiaphragmatic paralysis after block

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No